CLINICAL TRIAL: NCT03339856
Title: Selective Retina Therapy With Real-Time Feedback-Controlled Dosimetry for Treating Acute Idiopathic Central Serous Chorioretinopathy in Korean Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kim's Eye Hospital (Other)
Responsible Party: Principal Investigator, Jae Hui Kim, Principal Investigator, Kim's Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-116571-AB-N-01
Record Dates: First submitted 2017-11-06; First posted 2017-11-13 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2017-11

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients received selective retina therapy
  Interventions: Device: Selective retina therapy

INTERVENTIONS:
Device: Selective retina therapy — The selective retina therapy (SRT) is a laser treatment to the retina using the R:GEN device (Lutronic, Goyang-si, South Korea).
  Laser energy began at 80 µJ and was increased in 5-10 µJ intervals until the optimal energy delivery was confirmed by the RFD system. Following confirmation, the optimal laser energy was applied to fluorescein leakages. If the energy was indeed optimal at leakage points, laser shots were administered around the leakages. If the energy was not optimal at the leakage points, laser energy was again increased in 5-10 µJ increments until optimal energy delivery.

SUMMARY:
Selective retina therapy (SRT) selectively disrupts the retinal pigment epithelium (RPE) with minimal damage to the photoreceptors. Previous studies have shown SRT to be effective for resolving SRF, while causing only minimal collateral damage to the retina and vision.However, most patients included in prior studies had chronic CSC (≥3 months symptom duration) and SRT efficacy on acute CSC is not fully known.

The current study evaluated short-term treatment outcomes following SRT with real-time feedback-controlled dosimetry in Korean patients with acute idiopathic CSC.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is a disorder that is characterized by a localized serous detachment of the neurosensory retina in the posterior pole. Additionally, CSC is often self-limiting and spontaneous resolution of subretinal fluid (SRF) often occurs within several months. Although several treatment modalities (e.g., laser photocoagulation, photodynamic therapy, and anti-vascular endothelial growth factor [VEGF] therapy have been used in CSC patients, a consensus has not yet been reached on the optimal time for intervention.

Selective retina therapy (SRT) selectively disrupts the retinal pigment epithelium (RPE) with minimal damage to the photoreceptors. Previous studies have shown SRT to be effective for resolving SRF, while causing only minimal collateral damage to the retina and vision. However, most patients included in prior studies had chronic CSC (≥3 months symptom duration) and SRT efficacy on acute CSC is not fully known.

When treating CSC patients, it is generally recommended to follow-up several months without any intervention to identify spontaneous resolution of SRF. However, prompt treatment may be beneficial for some patients. For example, metamorphopsia or micropsia associated with CSC can greatly interfere with driving or with work when an occupation requires delicate procedures. Additionally, patients are often psychologically distressed by a CSC diagnosis and the accompanying decrease in vision-related quality of life. In these cases, prompt treatment to reduce SRF may relieve, at least in part, CSC symptoms and their related stress.

The current study evaluated short-term treatment outcomes following SRT with real-time feedback-controlled dosimetry in Korean patients with acute idiopathic CSC.

This study included patients who were diagnosed with treatment-naïve idiopathic CSC and were treated with SRT. The R:GEN device (Lutronic, Goyang-si, South Korea) was used to administer SRT. Inclusion criteria also included SRF involving the fovea (documented by optical coherence tomography [OCT] performed at initial presentation) and symptom duration shorter than 3 months. Patients were excluded from analyses if any of the following were true: (1) age > 55 years, (2) clinical or angiographic features suggestive of choroidal neovascularization, (3) OCT findings suggestive of type 1 neovascularization or polypoidal choroidal vasculopathy (e.g., double layer sign or fibrovascular pigment epithelial detachment), (4) history of macular laser photocoagulation, photodynamic therapy, or anti-VEGF therapy, or (5) history of exogenous corticosteroid treatment for a systemic disease (e.g., Cushing's syndrome or renal disease).

Examination, treatment, and follow-up All subjects underwent comprehensive ophthalmologic examinations, including best-corrected visual acuity (BCVA) measurement, slit-lamp biomicroscopy (90-diopter lens), fluorescein angiography (FAG), fundus photography, and spectral domain OCT (Spectralis HRA-OCT™, Heidelberg Engineering, Dossenheim, Germany or RS 3000™, Nidek Co., Ltd., Tokyo, Japan). Indocyanine green angiography using a confocal laser-scanning system (Spectralis HRA-OCT™) was performed at the discretion of each physician. A CSC diagnosis was based on FAG findings, in particular, evidence of a typical ink blot or smokestack leakage. A single examiner (J.H.K.) reviewed all FAG results.

All SRT was performed by a single physician (J.H.K.) using a Nd:YLF laser (wavelength of 257 nm, 15 micro pulses per spot, single micro pulse duration of 1.7 µs, pulse repetition rate of 100 Hz). Spot size was set at a diameter of 200 µm. Real-time feedback-controlled dosimetry (RFD) detects ultrasonic pressure waves generated by intracellular bubble formation and was used to determine optimal laser energy. Before applying laser energy to a leakage point, test shots were made immediately outside of the superior or inferior temporal arcade.

Optimal laser energy was determined based on real-time feedback system indications on the control panel. Laser energy began at 80 µJ and was increased in 5-10 µJ intervals until the optimal energy delivery was confirmed by the RFD system. Following confirmation, the optimal laser energy was applied to fluorescein leakages. If the energy was indeed optimal at leakage points, laser shots were administered around the leakages. If the energy was not optimal at the leakage points, laser energy was again increased in 5-10 µJ increments until optimal energy delivery, as confirmed by the RFD system. If the control panel indicated that excessive laser energy had been applied, the laser energy was decreased in 5-10 µJ increments until the optimal energy delivery was again achieved (confirmed by RFD system). The total number of laser shots delivered around fluorescein leakage points that were at or above the optimal laser energy were counted.

Patients had follow-up visits 1 and 3 months after SRT, at which BCVA was measured and OCT examination was performed. Central foveal thickness (CFT) was manually measured on OCT images and was defined as the distance between the RPE and the internal limiting membrane.

Outcome measures Both BCVA and CFT were measured at diagnosis, at 1 and 3 months following SRT, and at the final follow-up visit. The incidence of complete SRF resolution was estimated. Color fundus photographs taken at each follow-up visit also documented laser treatment and were used to check for the presence of visible laser spots. All BCVA measurements were converted to the logarithm of the minimum angle of resolution (logMAR) for data analyses.

Statistical analyses Statistical analyses were performed using a commercially available software package (SPSS v. 12.0 for Windows; SPSS Inc., Chicago, IL). Comparisons between BCVA and CFT measurements at different time points were performed using Wilcoxon signed-rank tests with a Bonferroni correction. Statistical significance was defined as P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with treatment-naïve idiopathic central serous chorioretinopathy

Exclusion Criteria:

* age > 55 years,
* Clinical or angiographic features suggestive of choroidal neovascularization
* Optical coherence tomography findings suggestive of type 1 neovascularization or polypoidal choroidal vasculopathy (e.g., double layer sign or fibrovascular pigment epithelial detachment).
* History of macular laser photocoagulation, photodynamic therapy, or anti-vascular-endothelial growth factor therapy.
* History of exogenous corticosteroid treatment for a systemic disease (e.g., Cushing's syndrome or renal disease).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Subretinal fluid | 3 months after treatment
  Presence or absence of subretinal fluid which identified based on optical coherence tomography images.

SECONDARY OUTCOMES:
Visual acuity | At diagnosis, at 1 month, and 3 months after treatment
  Changes in logarithm of minimal angle of resolution visual acuity during the follow-up, which measured using visual acuity chart.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim YJ, Lee YG, Lee DW, Kim JH. Selective Retina Therapy with Real-Time Feedback-Controlled Dosimetry for Treating Acute Idiopathic Central Serous Chorioretinopathy in Korean Patients. J Ophthalmol. 2018 Feb 6;2018:6027871. doi: 10.1155/2018/6027871. eCollection 2018. PMID 29545953